CLINICAL TRIAL: NCT04600687
Title: Comparison of the Ease of Swallowability of B/F/TAF Placebo Compared to DTG/ABC/3TC Placebo
Brief Title: B/F/TAF Ease of Swallowability Trial
Acronym: BEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, John E. McKinnon, MD, MSc, Senior Staff, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Gilead Study #CO-US-380-4657
Record Dates: First submitted 2019-04-02; First posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: HIV Infections
Keywords: HIV; adherence; tolerability
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to take the first placebo tablet and within 30 minutes then take the second placebo tablet. The participants will complete questionnaires prior to taking any placebo pill and after each dose.
Masking Description: Neither the participant nor the person administering the questionnaires will know which placebo tablet the patient has been randomized to receiving first prior to study enrollment. The allocation of which placebo tablet is first swallowed will be randomized in a block randomization design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): Participants will be enrolled in a single arm with a cross over design. Each participant will receive both placebo tablets about 30 minutes apart. Questionnaires will be completed prior to and after each placebo tablet is swallowed.
  Interventions: Other: Placebo tablets

INTERVENTIONS:
Other: Placebo tablets — Participants will take placebo tablets identical to the commercial versions of the two combination antiretroviral single tablet regimens of bictegravir/emtricitabine/tenofovir alanfenamide and dolutegravir/abacavir/lamivudine.

SUMMARY:
The trial will assess the tolerability and swallowability of a STR placebo of B/F/TAF as compared to DTG/ABC/3TC placebo STR in healthy individuals and HIV antiretroviral naïve patients. The study team will evaluate the ease of swallow and patient's tolerance of the medication formulation, an important, yet often overlooked aspect of ART adherence, with the potential for significant impact on patient's outcomes.

DETAILED DESCRIPTION:
The study will plan to recruit 50 volunteers who will be randomized to receive Placebo A (B/F/TAF) or Placebo B (DTG/ABC/3TC). Randomization will ensure that the patients will have equal opportunity to try either placebo tablet first to avoid bias. Randomization will be done by an investigator not evaluating or providing the questionnaires to the patient. Participants will complete a questionnaire regarding what medications they take and what factors they consider affect their ease to swallow pills or tablets. The participants will be administered one of the placebo tablet with the research investigator present and will complete a questionnaire immediately following the first placebo dose. A study timeout for 15-30 minutes will be done following completion of the questionnaires. After which, participants will take the second placebo tablet and complete the final questionnaires.

The primary comparison will be between the placebo tablets A and B for tolerability, ease of swallow and participant preference. The investigators estimate that the sample size needed to detect a difference of at least 1 point in a 5 point Likert scale will be 50 patients with a standard deviation of 2 points, with >90% power.

ELIGIBILITY:
Inclusion Criteria:

1. HIV seronegative or seropositive treatment naïve adult over 18 years of age, currently in stable condition, ambulatory and able to swallow tablets or pills.
2. Patients able to provide informed consent and remain in clinic for at least 2 hours.
3. Study participants able to complete the study questionnaires.
4. No known history of allergies to any of the placebo components.

Exclusion Criteria:

1. Patients with known dysphagia or motility disorders leading to difficulty swallowing liquids, food or medications.
2. Patients allergic to any component of the placebo tablets.
3. Children under the age of 18 years.
4. Adults unable to provide informed consent.
5. Female patients known to be pregnant.
6. HIV seropositive patients on antiretroviral therapy or with prior history of antiretroviral therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2019-05-08 (Actual); Study Completion 2020-10-10 (Actual)

PRIMARY OUTCOMES:
Comparison of the ease of swallowability and tolerability of two antiretroviral placebo tablets | One hour
  To evaluate the ease and tolerability of swallowing and tolerability of two antiretroviral placebo tablet representing Bictegravir/Emtricitabine/TAF (B/F/TAF) single tablet as compared to a placebo tablet representing Dolutegravir/Abacavir/Lamivudine (DTG/ABC/3TC) by Likert scale questionnaire assessment.

SECONDARY OUTCOMES:
Impact of pill/tablet size of two antiretroviral placebo tablets on acceptability for patients for adherence. | One hour
  To assess whether a smaller pill/tablet size is associated with better acceptance by patients by questionnaire.
Tablet characteristics that matter to patients for ease of swallow and for adherence | One hour
  To determine which particular tablet characteristic is more important as indicated by patients that affects their acceptance of a particular tablet or medication by questionnaire.
Patient's ease of swallow and medication preferences impact on medication adherence | One hour
  To assess patients' view on how pill/tablet size and ease of swallow impacts their medication adherence by questionnaire using a Likert scale.
How patient's cultural differences affect acceptability of pill/tablet size | One hour
  To determine if there are any cultural or ethnic differences in pill/tablet acceptance or ease of swallow.

CONTACTS AND LOCATIONS:
Overall Officials: John E. McKinnon, MD, MSc, Principal Investigator — Henry Ford Health System
Locations (1):
- John McKinnon, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided
After completion of the study and publication of the manuscript(s), the data will be made available for other researchers upon written request and review of the principal investigator.

REFERENCES:
- [Background] Bhosle M, Benner JS, Dekoven M, Shelton J. Difficult to swallow: patient preferences for alternative valproate pharmaceutical formulations. Patient Prefer Adherence. 2009 Nov 3;3:161-71. doi: 10.2147/ppa.s5691. PMID 19936158
- [Background] de Argila CM, Ponce J, Marquez E, Plazas MJ, Galvan J, Heras J, Porcel J. Acceptability of lansoprazole orally disintegrating tablets in patients with gastro-oesophageal reflux disease : ACEPTO study. Clin Drug Investig. 2007;27(11):765-70. doi: 10.2165/00044011-200727110-00003. PMID 17914895
- [Background] FDA. Size, Shape, and Other Physical Attributes of Generic Tablets and Capsules Guidance for Industry June 2015
- [Background] Fields J, Go JT, Schulze KS. Pill Properties that Cause Dysphagia and Treatment Failure. Curr Ther Res Clin Exp. 2015 Aug 20;77:79-82. doi: 10.1016/j.curtheres.2015.08.002. eCollection 2015 Dec. PMID 26543509
- [Background] Kakuda TN, Berckmans C, De Smedt G, Leemans R, Leopold L, Peeters M, Nijs S, Vyncke V, van Solingen-Ristea R, Hoetelmans RM. Single-dose pharmacokinetics of pediatric and adult formulations of etravirine and swallowability of the 200-mg tablet: results from three Phase 1 studies. Int J Clin Pharmacol Ther. 2013 Sep;51(9):725-37. doi: 10.5414/CP201770. PMID 23924679
- [Background] Nausieda PA, Pfeiffer RF, Tagliati M, Kastenholz KV, DeRoche C, Slevin JT. A multicenter, open-label, sequential study comparing preferences for carbidopa-levodopa orally disintegrating tablets and conventional tablets in subjects with Parkinson's disease. Clin Ther. 2005 Jan;27(1):58-63. doi: 10.1016/j.clinthera.2005.01.004. PMID 15763606
- [Background] Schiele JT, Quinzler R, Klimm HD, Pruszydlo MG, Haefeli WE. Difficulties swallowing solid oral dosage forms in a general practice population: prevalence, causes, and relationship to dosage forms. Eur J Clin Pharmacol. 2013 Apr;69(4):937-48. doi: 10.1007/s00228-012-1417-0. Epub 2012 Sep 29. PMID 23052416
- [Background] Singh JA. Facilitators and barriers to adherence to urate-lowering therapy in African-Americans with gout: a qualitative study. Arthritis Res Ther. 2014 Mar 29;16(2):R82. doi: 10.1186/ar4524. PMID 24678765